CLINICAL TRIAL: NCT05228821
Title: An Open Label, Single Arm, Multicenter Study to Evaluate the Effect of Voxelotor on Cerebral Blood Flow and Neurocognitive Function in Adolescents and Adults With Sickle Cell Disease
Brief Title: Voxelotor Brain Oxygenation and Neurocognitive Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study has been stopped due to Sponsor's business reasons. The termination is not a result of any safety concerns or change in the benefit-risk ratio.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBT440-043; C5341027 (Other: Alias Study Number)
Record Dates: First submitted 2022-01-10; First posted 2022-02-08 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Drug (Experimental): Generic Name: Voxelotor Dosage Form: tablet Dosage: 1500mg Frequency: QD Duration: 24 weeks
  Interventions: Drug: Voxelotor Oral Tablet

INTERVENTIONS:
Drug: Voxelotor Oral Tablet — During the Treatment Period, participants will receive 1500 mg of voxelotor once daily (administered as tablets) for 24 weeks in addition to ongoing current standard of care (SOC) treatment
  Other Names: Oxbryta

SUMMARY:
This is an open label, single arm multicenter trial to evaluate the effect of voxelotor treatment on cerebral blood flow (CBF) and neurocognitive function in adolescent and young adult participants (12-30 years of age) with sickle cell disease (SCD).

DETAILED DESCRIPTION:
Eligible participants will receive daily treatment with 1500 mg voxelotor for 24 weeks. During screening, at 12 and 24 weeks, participants will undergo an MRI for evaluation of cerebral blood flow and oxygen extraction fraction as well as NIH toolbox testing for evaluation of executive function, processing speed, and nonexecutive function.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants with confirmed diagnosis of SCD with HbSS or Hbβ0 thalassemia genotype. Documentation of SCD genotype is required and may be based on documented history of laboratory testing or confirmed by laboratory testing during Screening.
2. Aged 12 to 30 years.
3. Screening Hb level ≥ 5.5 and ≤ 10.5 g/dL.
4. Must meet site-specific compliance requirements for a diagnostic MRI scan.
5. Able to answer NIH Toolbox Module questions in English
6. If participant is receiving hydroxyurea (HU) they must have been on a stable dose for at least 90 days prior to signing the ICF/AF, with no dose modifications or initiation of HU planned or anticipated by the Investigator.
7. If participant is receiving erythropoiesis-stimulating agents (ESAs) they must have been on a stable dose for at least 12 weeks before enrollment with no dose modifications planned or anticipated by the Investigator.
8. Participants, who if female and of child-bearing potential, agree to use highly effective methods of contraception from study start to 30 days after the last dose of study drug and who if male, agree to use barrier methods of contraception and refrain from donating sperm from study start to 30 days after the last dose of study drug.
9. Females of child-bearing potential must have a negative pregnancy test before the administration of study drug.
10. Written informed consent (≥ 18 years) or parental/guardian consent and participant assent (≥ 12-17 years) per Institutional Review Board (IRB) policy and requirements, consistent with ICH guidelines.
11. Capable of complying with the requirements and restrictions in the protocol, and willing to participate in the study.

Exclusion Criteria:

1. History of overt stroke including hemorrhagic stroke, transient ischemic attacks, or spinal cord injury.
2. Grade 4 vasculopathy defined as moderate stenosis (50% to 69%) in more than 2 major cerebral arteries or severe stenosis (> 70%) in any major cerebral artery.
3. Non-MRI compatible metal hardware and/or metal braces.
4. Congenital brain malformation, previously diagnosed severe developmental disability (eg autism and/or intelligence quotient [IQ] <60, and/or severe attention deficit hyperactivity disorder [ADHD]), or impairment that would prevent the use of a computer tablet.
5. Participant is taking or has received voxelotor (Oxbryta®) within 90 days prior to the Screening Visit.
6. Participant is taking or has received crizanlizumab (Adakveo®) within 90 days prior to the Screening Visit.
7. Vaso-occlusive event requiring intravenous opioids within 28 days prior to Day 1.
8. Red blood cell (RBC) transfusion within 3 months before initiation of study drug or receives scheduled RBC transfusion therapy (also termed chronic, prophylactic, or preventive transfusion).
9. Surgery within 8 weeks before Day 1 or planned elective surgery during the study.
10. Anemia due to bone marrow failure (eg, myelodysplasia).
11. Absolute reticulocyte count (ARC) < 100 × 10^9/L.
12. Screening alanine aminotransferase or aspartate aminotransferase > 4× upper limit of normal (ULN).
13. Severe renal dysfunction (estimated glomerular filtration rate [eGFR] <45 mL/min/1.73 m^2) or on chronic dialysis.
14. Clinically significant bacterial, fungal, parasitic, or viral infection which requires therapy

    1. Acute bacterial infection requiring antibiotic use should delay Screening/enrollment until the course of antibiotic therapy has been completed.
    2. Known active hepatitis A, B, or C or are known to be human immunodeficiency virus (HIV) positive.
15. Symptomatic coronavirus disease of 2019 (COVID-19) infection.
16. Females who are breast-feeding or pregnant.
17. History of hematopoietic stem cell transplant or gene therapy.
18. Participants taking concomitant medications such as sensitive CYP3A4 substrates with a narrow therapeutic range, or strong CYP3A4 inducers.
19. Participated in another clinical trial of an investigational product (or medical device) within 30 days or 5 half-lives of date of informed consent, whichever is longer, or is currently participating in another trial of an investigational product (or medical device).
20. Medical, psychological, or behavioral condition that, in the opinion of the Investigator, would confound or interfere with evaluation of safety and/or efficacy of the study drug, prevent compliance with the study protocol; preclude informed consent; or render the participant unable/unlikely to comply with the study procedures (particularly the MRI scan).

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Change in CBF | Baseline to Week 24
  Change from Baseline in CBF through Week 24 measured by magnetic resonance imaging (MRI) using pseudo-continuous arterial spin labeling (pCASL).

SECONDARY OUTCOMES:
Change in executive functioning. | Baseline to Week 24
  Change from Baseline through Week 24 in the executive cognitive abilities composite score (using Dimensional Change Card Sort Test, Flanker Inhibitory Control and Attention Test, and List Sorting Test) as assessed by the National Institutes of Health Toolbox Cognition Module.
Change in processing speed | Baseline to Week 24
  Change from Baseline through Week 24 in processing speed (using Pattern Comparison Test) as assessed by the NIH Toolbox Cognition Module
Change in nonexecutive functioning | Baseline to Week 24
  Change from Baseline through Week 24 in nonexecutive cognitive abilities composite score (using Picture Vocabulary Test, Oral Reading Recognition Test, and Picture Sequence Memory Test) as assessed by the NIH Toolbox Cognition Module.

OTHER OUTCOMES:
Change in Hb and hemolysis over time | Baseline to week 24
  Change and percent change from Baseline through Week 24 in hemolysis measures, including unconjugated bilirubin, absolute reticulocyte, % reticulocytes, and lactate dehydrogenase (LDH).
Change in cerebral dynamics | Baseline to week 24
  Change from baseline through Week 24 in cerebral blood flow, oxygen extraction, and oxygen metabolism as measured by diffusion correlation spectroscopy (DCS)/frequency domain near infrared spectroscopy (FDNIRS) (if available)
  Correlation of cerebral hemodynamics measured by DCS/FDNIRS (if available) and cerebral hemodynamics measured by MRI.
Change in global OEF as measured using T2-Relaxation-Under-Spin-Tagging (TRUST) | Baseline to week 24
  Change from Baseline to Week 24 in global OEF as measured using TRUST (if available)).
Change in regional CBF within the grey matter | Baseline to Week 24
  Change from Baseline through Week 24 in regional CBF within the grey matter.
Change in regional CBF within the white matter | Baseline to Week 24
  Change in HRQOL scores using:
  Change from Baseline through Week 24 in regional CBF within the white matter
Change in regional OEF as measured using ASE (If available) | Baseline to week 24
  Change from Baseline to Week 24 in regional OEF as measured using ASE (if available)
Correlation between changes from Baseline in CBF (MRI and DCS/FDNIRS) | Baseline to Week 24
  Correlation between changes from Baseline in CBF (MRI and DCS/FDNIRS) and changes from Baseline in Hb levels
Correlation of changes from Baseline in OEF (MRI and DCS/FDNIRS) | Baseline to Week 24
  Correlation of changes from Baseline in OEF (MRI and DCS/FDNIRS) and changes from Baseline in Hb levels
Correlation of change from Baseline in Hb | Baseline to Week 24
  Correlation of change from Baseline in Hb and change from Baseline in executive abilities composite score
Change in HRQOL scores | Baseline to Week 24
  Change in HRQOL scores using Patient Global Impression of Severity (PGI-S)
Change in HRQOL scores using Clinician Global Impression of Severity. | Baseline to Week 24
  Change in HRQOL scores using Clinician Global Impression of Severity (CGI-S)
Incidence and severity of treatment-emergent AEs (TEAEs) | Baseline to Week 24
  Incidence and severity of treatment-emergent AEs (TEAEs) baseline through week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - The Children's Hospital at Montefiore, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-043